CLINICAL TRIAL: NCT00766324
Title: A Phase II Study of PHA-739358 in Patients With Metastatic Hormone Refractory Prostate Cancer
Brief Title: PHA-739358 for Treatment of Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AURA-6202-007
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Metastatic Hormone Refractory Prostate Cancer
MeSH Terms: interventions — danusertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: PHA-739358
- B (Experimental)
  Interventions: Drug: PHA-739358

INTERVENTIONS:
Drug: PHA-739358 — 6-hr IV infusion weekly for 3 consecutive weeks in a 4-week cycle
  Arms: A
Drug: PHA-739358 — 24-hr IV infusion every 2 weeks in a 4-week cycle
  Arms: B

SUMMARY:
To assess the antitumor activity of PHA-739358 administered as IV infusion according to two different dose schedules in metastatic HRPC patients progressing on standard, docetaxel-based 1st-line chemotherapy for HRPC based on PSA response, and to select the best dose schedule for further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic hormone refractory prostate cancer progressing after docetaxel based therapy
* Adequate bone marrow, liver and kidney function

Exclusion Criteria:

* More than one prior chemotherapy line
* Uncontrolled hypertension
* Brain or leptomeningeal disease
* Myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident in the previous 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
PSA response rate defined according to the recommendations from the Prostate-Specific Antigen Working Group | within the first three months of treatment

SECONDARY OUTCOMES:
Objective Response Rate, Progression Free Survival, additional PSA based endpoints, clinical benefit | all cycles
Overall safety profile | all cycles

CONTACTS AND LOCATIONS:
Locations (1):
- Nerviano Medical Sciences. Clinical Research Dept., Nerviano, Milano, Italy